CLINICAL TRIAL: NCT01394614
Title: Risk of Narcolepsy Associated With Administration of Inactivated Adjuvanted (AS03) A/H1N1 Pandemic Influenza Vaccine in Quebec
Brief Title: Risk of Narcolepsy Associated With Administration of H1N1 Vaccine
Status: Completed | Type: Observational
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Jacques Montplaisir, Director of the Sleep Clinic, Sacre-Coeur Hospital, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Other Study IDs: Narco-H1N1
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Narcolepsy
Keywords: Cataplexy; MSLT; Hypocretin; HLA typing; Polysomnography; A/H1N1 vaccine
MeSH Terms: conditions — Narcolepsy; Cataplexy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — HLA typing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Narcoleptics exposed to A/H1N1 vaccine: Adjuvanted (ASO3) A/H1N1 pandemic vaccine
  Interventions: Biological: A/H1N1 vaccine
- Narcoleptics unexposed to A/H1N1 vaccine: Narcoleptic subjects who were unexposed (non-vaccinated or vaccinated after onset) to adjuvanted (ASO3) A/H1N1 pandemic vaccine.

INTERVENTIONS:
Biological: A/H1N1 vaccine — Verify if exposure to Arepanrix vaccine increase risk of developing narcolepsy in 16 weeks post-vaccination.
  Other Names: Arepanrix vaccine
  Groups: Narcoleptics exposed to A/H1N1 vaccine

SUMMARY:
The goal of the study is to assess the risk of occurrence of narcolepsy following the administration of inactivated (AS03) adjuvanted A/H1N1 pandemic influenza vaccine in the province of Quebec, Canada, using different case definitions and time intervals to disease onset, while controlling for potential confounding variables such as age, gender, season and, when possible, A/H1N1 pandemic influenza infection. Another aim is to describe the epidemiology and clinical features of narcolepsy cases with onset during the period January 1st, 2009 to December 31, 2010 in the population of Quebec.

DETAILED DESCRIPTION:
This study aims to describe the epidemiological and clinical characteristics of cases of narcolepsy which occurred in Quebec during the period 1 January 2009 to December 31, 2010 and to assess the risk of developing narcolepsy associated with the vaccine against influenza A/H1N1. The study will last about six months. Based on the prevalence of narcolepsy, an estimated 100 people who developed symptoms of narcolepsy between January 1st, 2009 and December 31, 2010 will participate in this study at the sleep clinic of the Sacré-Coeur Hospital in Montreal.

Narcolepsy is primarily characterized by the presence of excessive daytime sleepiness (EDS) and cataplexy. EDS occurs daily and is usually the most disabling symptom of narcolepsy. Cataplexy consists of a sudden drop of muscle tone triggered by strong and sudden emotions such as laughter, anger and surprise. Cataplexy is the most specific symptom of narcolepsy but it is not present in every patient especially at disease onset. Two other auxiliary symptoms are sleep paralysis and hypnagogic hallucinations either at sleep onset or upon awakening during the night or in the morning. They are present in approximately two thirds of narcoleptic patients especially in the younger individuals during the early stage of narcolepsy. Narcolepsy is associated with an absence or low level of hypocretin1 peptide in the cerebrospinal fluid (CSF).

Narcolepsy with cataplexy can be diagnosed purely on clinical grounds but this diagnosis should whenever possible be confirmed by night-time polysomnography (PSG) followed by the daytime multiple sleep latency test (MSLT). Sleep latency on the MSLT should be inferior or equal to 8 minutes with the presence of two or more sleep onset REM periods (SOREMPs). Human leukocyte antigen (HLA) typing of patients with narcolepsy-cataplexy almost always shows the presence of HLA DQB1*0602. Finally, measuring CSF level of hypocretin-1 is specific and sensitive for the diagnosis of narcolepsy with cataplexy.

Cases of narcolepsy following administration of A/H1N1 pandemic vaccines have been reported in Sweden, Finland, France and Canada. The majority of reports have shown a temporal association with inactivated (AS03) adjuvanted A/H1N1 vaccines. These cases had some common features: severe sleepiness and presence of cataplexy, abrupt onset and rapid evolution, presence of HLA DBQ1*0602 marker, very low CSF hypocretin-1, and positive MSLT test. At the request of the European Medicines Agency (EMA), a series of investigations have been considered by GlaxoSmithKline Biologicals, including one in Quebec. In this province, following the report of four cases of narcolepsy with cataplexy potentially associated with administration of Arepanrix, our research team was contacted both by federal and provincial public health authorities to evaluate the possibility of an independent investigation.

A retrospective cohort study is proposed. The existence of a comprehensive influenza immunization registry in Quebec allows a precise identification of the cohort of exposed subjects, by age and gender. Exposed subjects will be followed from the time of vaccine administration (first dose of inactivated AS03 A/H1N1 pandemic vaccine) as recorded in the immunization registry. The size of non-exposed subjects by gender- and age-specific categories will be estimated from the number in census data (a more accurate source than provincial health insurance data) minus the number in the influenza immunization registry. Pseudo-dates of vaccine administration will be generated for non-exposed subjects based on the distribution of dates of vaccinated subjects. Non-exposed subjects will be followed from the pseudo-date of vaccine administration.

All neurologists, pulmonologists, neuro-pediatricians and child psychiatrists practicing in the province of Quebec will be contacted and asked to report confirmed or suspected cases of narcolepsy with onset during the period from January1st, 2009 to December 31, 2010. Patients will be contacted by their physicians and invited to call the sleep center to participate in a study of newly diagnosed cases of narcolepsy. They will then undergo a brief screening telephone questionnaire. At this point, if they meet the minimum criteria of narcolepsy, they will be asked if they agree to participate in the study. The study includes, at first, signing a consent form and completing a questionnaire.

The questionnaire includes questions on demographics, medical history, medications, and detailed questions about symptoms of narcolepsy. In children, the information will be based on parental responses. A physician specializing in sleep medicine will call the participant to review the questionnaire with him and will propose a series of tests at the sleep laboratory of the 'Hôpital du Sacré-Coeur de Montréal', including nocturnal polysomnography, MSLT test, blood sampling (for HLA typing) and, lumbar puncture (for hypocretin measurements). Patients will sign a second consent form on site at 'Hôpital du Sacré-Coeur de Montréal' if they agree to participate in that second portion of the study. Monitoring of subjects during the study will be done under the supervision of Dr. Jacques Montplaisir, MD, PhD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with symptoms of narcolepsy with onset during the period between January 1st, 2009 and December 31, 2010.

Exclusion Criteria:

* Subjects younger than 6 months of age

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes persons more than 6 months of age residing in the province of Quebec.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Montplaisir, MD, PhD, Principal Investigator — Sacre-Coeur Hospital
Locations (1):
- Sacre-Coeur Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Montplaisir J, Petit D, Quinn MJ, Ouakki M, Deceuninck G, Desautels A, Mignot E, De Wals P. Risk of narcolepsy associated with inactivated adjuvanted (AS03) A/H1N1 (2009) pandemic influenza vaccine in Quebec. PLoS One. 2014 Sep 29;9(9):e108489. doi: 10.1371/journal.pone.0108489. eCollection 2014. PMID 25264897

RESULTS

PARTICIPANT FLOW:
Groups:
- Narcoleptic Subjects Exposed to Vaccine: Exposed narcoleptic subjects (vaccinated and onset of narcolepsy is after vaccine administration)
- Unexposed Narcoleptic Subjects: Unexposed narcoleptic subjects (not vaccinated or vaccinated after the onset of symptoms)
Period: Overall Study
Arm/Group | Narcoleptic Subjects Exposed to Vaccine | Unexposed Narcoleptic Subjects
Started | 8 | 16
Completed | 8 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Exposed Narcoleptic Subjects: Exposed (vaccinated and onset of narcolepsy is after vaccine administration) narcoleptic subjects to adjuvanted A/H1N1 vaccine
- Unexposed Narcoleptic Subjects: Unexposed (non-vaccinated or vaccinated after onset of symptoms) narcoleptic subjects to adjuvanted A/H1N1 vaccine
- Total: Total of all reporting groups
Arm/Group | Exposed Narcoleptic Subjects | Unexposed Narcoleptic Subjects | Total
Number analyzed (Participants) | 8 | 16 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 7 | 13
  Between 18 and 65 years | 2 | 9 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 19.9 [6 to 50] | 26.1 [8 to 55] | 24.0 [6 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 2 | 10 | 12
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 16 | 24

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Narcolepsy Among Narcoleptic Subjects Exposed or Unexposed to Vaccine
Description: Incidence rates will be computed by comparing narcolepsy incidence rates in exposed and non-exposed subjects. Comparison of narcolepsy incidence rates in the period prior to vaccine administration and pseudo-vaccine administration will be used to test the comparability of exposed and non-exposed group.
Time Frame: Narcolepsy onset during the 16-week post-vaccination period.
Measure: Number; unit: events per 100,000 person-years
Groups:
- Exposed Narcoleptic Subjects: Exposed (vaccinated and onset of narcolepsy is post-vaccination) narcoleptic subjects
  Intervention: Adjuvanted (ASO3) A/H1N1 pandemic vaccine Arepanrix.
- Unexposed Narcoleptic Subjects: Unexposed narcoleptic subjects (non-vaccinated or vaccinated after onset of symptoms)
Arm/Group | Exposed Narcoleptic Subjects | Unexposed Narcoleptic Subjects
Number analyzed (Participants) | 8 | 16
events per 100,000 person-years | 0.52 | 0.11
Statistical Analysis 1: Comparison: Exposed Narcoleptic Subjects vs Unexposed Narcoleptic Subjects; Test type: Superiority or Other; Incidence-rate difference = 0.41 — Difference between the incidence rate of exposed-to-vaccine cases (0.52) and that of unexposed cases (0.11) is 0.41 per 100,000 persons-years
Statistical Analysis 2: Comparison: Exposed Narcoleptic Subjects vs Unexposed Narcoleptic Subjects; Test type: Superiority or Other; Risk Ratio (RR) = 4.32, 95% CI 2-sided [1.5 to 11.12] — Risk of developing narcolepsy if exposed to H1N1 vaccination (using the 16-week post-vaccination period as reference)

ADVERSE EVENTS:
Time Frame: Adverse Events were not reported since this was a retrospective study (only onset of narcolepsy, which is the main outcome, was reported)
Groups:
- Exposed Narcoleptic Subjects: Exposed narcoleptic subjects (vaccinated and onset of narcolepsy is post-vaccination)
  Intervention: Adjuvanted (ASO3) A/H1N1 pandemic vaccine (Arepanrix)
Arm/Group | Exposed Narcoleptic Subjects | Unexposed Narcoleptic Subjects
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Small number of subjects; Impossibility to completely exclude a confounding effect of the A/H1N1 virus infection itself.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No